CLINICAL TRIAL: NCT05206630
Title: An Ancillary Cluster-Randomized Trial of Embedded Physical Therapy for Chronic Low Back Pain
Brief Title: ED Physical Therapy for Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Howard Kim, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00213134
Record Dates: First submitted 2022-01-11; First posted 2022-01-25 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Low Back Pain
Keywords: low back pain; chronic; physical therapy; emergency department; functioning; disability; opioid
MeSH Terms: conditions — Low Back Pain; Bronchiolitis Obliterans Syndrome; Emergencies

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Embedded ED Physical Therapy (Experimental): An ED physical therapist will be embedded with the primary treatment team to evaluate patients presenting with low back pain at the beginning of the overall treatment course. The physical therapist will utilize a clinical protocol that matches the patient's history and exam findings to an appropriate treatment classification consisting of directional preference exercises, manual traction, stabilization exercises, non-thrust manipulation/mobilization, and/or psychologically informed rehabilitation. The embedded PT intervention will supplement any usual care performed by the treating physician.
  Interventions: Other: ED Physical Therapy
- Usual Care (No Intervention): Usual care consists of any ED testing or treatment not involving an ED physical therapist in accordance with the treating physician's usual and customary practice. This could include diagnostic imaging, patient education and reassurance, and administration and/or prescribing of analgesic medications.

INTERVENTIONS:
Other: ED Physical Therapy — All ED Physical Therapy treatment classifications involve a combination of exercise, range of motion, education, prognostic guidance, and reassurance. Patients are provided with an individualized home exercise plan based on their matched treatment classification and/or active rest.
  Arms: Embedded ED Physical Therapy

SUMMARY:
Emergency department (ED)-initiated physical therapy is a rapidly growing resource and represents a promising treatment approach to low back pain. This clinical trial will evaluate an innovative model of an emergency department "embedded" physical therapist to treat patients with chronic low back pain, with a focus on improving patient functioning and reducing opioid use.

DETAILED DESCRIPTION:
This trial is ancillary to an ongoing single-center physician-randomized trial of an embedded physical therapy intervention versus usual care in ED patients with acute low back pain (NEED-PT, NCT04921449), comparing a primary outcome of pain-related functioning and a secondary outcome of opioid use at three months. The main trial aims to enroll up to 360 participants with acute low back pain, defined as ≤ 30 days in duration and no history of lumber surgery or chronic low back pain. Using the same procedures and physician-randomization assignments as the main trial, this ancillary trial will enroll an additional 200 participants with chronic low back pain (i.e. non-acute low back pain) in order to obtain initial point estimates for the outcomes of interest and assess participant enrollment and retention rates in this population. The ancillary trial's sample size of 200 participants is an estimate of patient accrual over the anticipated remaining duration of the main trial (i.e., there is not a separate power calculation for this ancillary trial given its exploratory nature), and the actual number accrued may differ depending on the main trial's actual end date.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Low back pain (originating between 12th rib and buttocks)
* Evaluated by a physician randomized to either study arm
* Evaluated when ED physical therapy is available (e.g., Mon-Fri, 8am-4pm)
* Likely to be discharged home (based on physician assessment)
* Ability to complete follow-up data collection electronically or by telephone
* English-speaking

Exclusion Criteria:

* Enrollment in the main trial (NEED-PT, NCT04921449)
* Serious red-flag signs/symptoms (bladder/bowel incontinence, saddle anesthesia, debilitating motor weakness)
* Obvious non-musculoskeletal etiology for low back pain (e.g., shingles, kidney stone)
* Other concomitant injuries or pain (e.g., closed head injury, shoulder pain)
* Unable to ambulate at baseline
* Known pregnancy, under police custody, unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2024-10-03 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
PROMIS Pain Interference (PROMIS-PI) | Three months after the index ED visit.
  PROMIS-PI measures the self-reported consequences of pain on relevant aspects of a person's life, including social, cognitive, emotional, physical, and recreational activities. The investigators will use the computer-adaptive format to minimize respondent burden. Scores are standardized to the general U.S. population, with a score of 50 representing the population mean. The time frame of interest for the PROMIS-PI is "in the past 7 days," meaning that participants provide responses based on their symptoms over the last week.

SECONDARY OUTCOMES:
Modified Oswestry Disability Index (ODI) | Three months after the index ED visit.
  The ODI contains 10 questions relating to low back pain intensity, personal care, lifting, walking, sitting, standing, sleeping, social life, traveling, and employment/homemaking. The ODI score ranges from zero (no disability) to 100 (maximum disability). The time frame of interest for the ODI is "today," meaning that participants provide responses based on their current symptoms on the day of survey response. The modified ODI replaces an item from the original ODI pertaining to sex life with a new item pertaining to employment/homemaking.
Patient-Reported Opioid Use in Last 24 Hours | Three months after the index ED visit.
  Patient-reported opioid use will be collected using a customized instrument assessing whether participants have taken any opioid medication in the last 24 hours (binary yes/no). The 24-hour timeframe was selected to maximize accuracy in patient recall and has been used previously. In brief, opioid medications are listed by brand and generic names; a "yes" response to any medication triggers an additional query asking the participant to specify the medication dose (e.g., oxycodone 10mg) and quantity (e.g., four pills), allowing for standardization by morphine milligram equivalents.

OTHER OUTCOMES:
Opioid Prescription Filling | Three months after the index ED visit.
  Opioid prescription filling data will be queried in the state prescription monitoring database.
Patient-Reported Prescription Analgesic Use in Last 24 Hours | Three months after the index ED visit.
  Patient-reported prescription analgesic use will be collected using the same customized instrument described above for opioid use. Prescription analgesics include the following: opioids, benzodiazepines, skeletal muscle relaxants, and gabapentinoids.
Prescription Analgesic Filling | Three months after the index ED visit.
  Prescription analgesic filling data will be queried in the state prescription drug monitoring database. Prescription analgesics include opioids, benzodiazepines, skeletal muscle relaxants, and gabapentinoids.
Numeric Pain Rating Scale (NPRS) | Three months after the index ED visit.
  The NPRS measures pain intensity from 0 to 10 (higher score indicates higher intensity) and is easily understood by laypersons, clinicians, and researchers. The investigators will assess a single item relating to average pain intensity over the last 24 hours.
Global Rating of Change (GROC) | Three months after the index ED visit.
  The GROC is a single-item survey used to evaluate overall recovery from low back pain from "the time that you began having pain until now." Responses are provided on a 15-point Likert scale ranging from "a very great deal worse" to "a very great deal better" (higher scores indicate better outcome).
Pain Catastrophizing Scale (PCS-4) | Three months after the index ED visit.
  The original PCS is a 13-item survey measuring the degree to which an individual catastrophizes in response to pain. PCS scores correlate closely with pain intensity and disability over time; higher PCS scores are associated with progression from acute to chronic pain. The investigators will utilize the brief 4-item PCS measure containing original items 3, 6, 8, and 11 (total score range 0-16, higher score indicates higher catastrophizing).
Pain Self-Efficacy Questionnaire (PSEQ-4) | Three months after the index ED visit.
  The original PSEQ is a 10-item survey measuring the confidence with which individuals can do things despite pain. The investigators will utilize the brief 4-item PSEQ measure containing original items 4, 6, 8, and 9 (total score range 0-24, higher score indicates higher confidence).
Advanced Healthcare Resource Utilization | Three months after the index ED visit.
  The investigators will assess the proportion of participants who utilized any advanced healthcare resources for low back pain after their index ED visit, defined as advanced imaging (e.g., magnetic resonance imaging) or procedures/surgery (e.g., epidural steroid injection, lumbar discectomy).
ED Diagnostic Imaging Utilization | Index ED 1 day visit.
  The investigators will assess the proportion of ED visits in which any diagnostic imaging of the lower back was performed, including plain radiography, computed tomography, or magnetic resonance imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Howard S Kim, MD MS, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No